CLINICAL TRIAL: NCT04758520
Title: Motor Rehabilitation of the Shoulder Complex After Orthopaedic Injury or Surgery Because of Work Accidents: a Pilot Study.
Brief Title: Usability and Acceptance of a New Robotic Exoskeleton for Shoulder Rehabilitation
Acronym: CRMINAIL08
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istituto Nazionale Assicurazione contro gli Infortuni sul Lavoro (Other)
Collaborators: Istituto Italiano di Tecnologia (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: CRMINAIL08
Record Dates: First submitted 2021-02-09; First posted 2021-02-17 (Actual); Last update posted 2022-03-31 (Actual); Status verified 2022-03

CONDITIONS: Shoulder Injuries and Disorders
Keywords: Adult; Deseases/musculoskeletal; Feasibility Studies; Humans; Occupational Therapy; Rehabilitation Research; Robotics; Shoulder Joint / therapy; Upper arm/therapy; Wearable devices
MeSH Terms: conditions — Shoulder Injuries; Disease

STUDY DESIGN:
Intervention Model Description: Single Group Assignment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental (Experimental): Six subjects are involved in a single session of upper limb robotic-assisted therapy lasting about 3 hours and including:
  * passive mobilization of patient's upper arm along elementary shoulder movements:shoulder flexion/extension, adduction/ abduction in the frontal plane, horizontal adduction/ abduction, intra/extrarotation (Passive Mode);
  * passive mobilization of patient's upper arm along complex trajectories recorded from manual mobilization of the therapist (Learn&Replay Mode);
  * active mobilization, performed by the patient during rehabilitative functional tasks, relying only on gravity and friction compensations and tuneable assistance from the exoskeleton (Transparency Mode).
  Interventions: Device: FLOAT upper limb exoskeleton

INTERVENTIONS:
Device: FLOAT upper limb exoskeleton — The FLOAT device is composed by a wearable exoskeleton assembled on a poly-articulated arm that, in turn, is mounted on a support base with unlockable wheels. The exoskeleton includes 5 motors arranged in a way that, when generating movement, ensures the optimal involvement of all the articulations of the shoulder complex, particularly the glenohumeral and the scapulothoracic joints. According to the chosen modality of use of the exoskeleton, the device allows patient's passive or active-assisted mobilization. The poly-articulated arm supporting the exoskeleton is capable to compensate exoskeleton weight in every configuration and, if configured appropriately, permits exoskeleton use both in seated and standing positions. The support base of the device has unlockable wheels that, if unlocked, permit the free movement of the patient in the workspace, enabling the performance of more complex functional activities while assisted by the exoskeleton.

SUMMARY:
The purpose of this pilot study is to validate the safety, reliability and usability of FLOAT medical device, a prototypal robotic system for the rehabilitation of the shoulder, designed and developed in the Rehab Technologies IIT-INAIL Lab to fulfil the needs orthopaedic conditions. The acceptance from patients and therapists will be assessed after a single session of robotic therapy in a sample of injured workers suffering from post-traumatic or post-surgical shoulder disorders.

DETAILED DESCRIPTION:
This study aims to:

1. Test the safety and reliability of the FLOAT device for delivering post-acute motor and functional rehabilitation of patients with orthopaedic shoulder dysfunction.
2. Assess the three different modalities of utilization of the exoskeleton (Passive Mode, Learn&Repeat Mode, Transparency Mode).
3. Evaluate the usability of the device in terms of comfort, adaptability to different patients' anthropometrics, general functioning and overall satisfaction.

Six injured workers with shoulder post-traumatic and post-operative dysfunction will be enrolled in a single testing session at the INAIL Rehabilitation Center in Volterra. Pilot testing of FLOAT device will focus mainly on the feasibility of implementing the multiple operating modes of the new device, recording patients and therapist's feedback. The session will last about 3 hours and all exercises will be administered by a trained physical therapist supported by a member of the engineering team.

For Aim 1, Safety and Reliability of the device will be evaluated in terms of the number of adverse events and malfunctions occurring during the study session.

For Aim 2, each modality will be assessed by means of the Numeric Pain Rating Scale (NPRS), The Borg CR10 Scale Perceived Exertion (only for the Transparent mode) and ad-hoc clinician-generated questionnaires for both patients and therapists.

For aim 3, patient and therapist's general evaluation about usability will be detected through a final ad-hoc questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Height between 160 and 185 cm;
* Distance between the shoulder joint center and the sagittal plane between 156 and 197 mm;
* Shoulder joint center to wall distance between 82 and 142 mm
* Maximum shoulter radius: 120 mm
* Distance between the shoulder joint center and the elbow joint center between 250 and 303 mm
* Time from acute event ≥ 60 days
* Right shoulder joint disfunction after orthopaedic injury or surgery as a result of work accidents
* Post-immobilization phase
* At least 80° shoulder passive flexion and 45° shoulder passive abduction
* Pain intensity on movement < 6 NRS;

Exclusion Criteria:

* Glenohumeral joint instability
* Shoulder Prosthetic implants
* Upper arm sensorimotor deficits
* Chronic inflammatory disorder involving upper arm joints
* Pseudoarthrosis of the proximal humerus fractures
* Spinal fractures within the last 3 months
* Open skin at the level of the patient-device interface
* Current or prior history of malignancy
* Pregnancy or breast feeding

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2020-11-20 (Actual); Primary Completion 2022-02-21 (Actual); Study Completion 2022-02-21 (Actual)

PRIMARY OUTCOMES:
Number of adverse events | 1 year
  The physiotherapist is required to report any adverse events occurring during the study in regard to the use of FLOAT, for the purpose of evaluating the safety of the device
Number of device malfunctions | 1 year
  The physiotherapist is required to report any malfunctions occurring during the study in regard to the use of FLOAT, for the purpose of evaluating the reliability of the device

SECONDARY OUTCOMES:
Numeric Pain Rating Scale (NPRS) | 1 year
  NPRS is an 11-point scale for patient self-reporting of pain, with 0 being "no pain" and 10 being "the worst pain imaginable"; It will be administered after each series of joint mobilization exercises.
The Borg Category-Ratio Scale (CR-10) | 1 year
  The Borg CR10 Scale is a tool for estimating effort and exertion, breathlessness, and fatigue during physical work, with rating ranges from 0 (nothing at all) to 10 (extremely strong).
  It will be administered after each series of functional tasks in transparent mode
Ad-hoc questionnaires for the patient, one for each of the three modalities (for a total amount of 3 questionnaires) | After the completion of the testing session with each of the three modalities
  Clinician-generated questionnaire to investigate patients' impressions about the physical interaction with the robotic device using the specific modality. Each questionnaire consists of a series of items with 5-point rating scale (1= not at all, 5=very well)
Ad-hoc questionnaires for the therapist, one for each of the three modalities (for a total amount of 3 questionnaires) | 1 year
  Clinician-generated questionnaire to investigate therapist's impressions about the usability and efficiency the robotic device using the specific modality. It will be administered after the completion of the testing session with each of the three modalities. Each questionnaire consists of a series of items with 5-point rating scale (1=not at all, 5=very well)
Ad-hoc questionnaire for the patient (final evaluation) | 1 year (at the end of the study)
  Clinician-generated questionnaire to investigate patients' general evaluation about FLOAT usability. The questionnaire consists of a series of items with 5-point rating scale (1=not at all, 5=very well)
Ad-hoc questionnaire for the therapist (final evaluation) | 1 year (at the end of the study)
  Clinician-generated questionnaire to investigate therapists' general evaluation about FLOAT usability. The questionnaire consists of a series of items with 5-point rating scale (1=not at all, 5=very well)

CONTACTS AND LOCATIONS:
Overall Officials: Elisa Taglione, MD, Principal Investigator — Istituto Nazionale Assicurazione contro gli Infortuni sul Lavoro
Locations (1):
- INAIL - Centro di Riabilitazione Motoria di Volterra, Volterra, Pisa, Italy

IPD SHARING:
Plan to Share IPD: No